CLINICAL TRIAL: NCT05290376
Title: Clinical Evaluation of RTX Locator Attachments for Implant-supported Mandibular Complete Overdenture Using Two Loading Protocols
Brief Title: Clinical Evaluation of RTX Locator Attachments for Implant-supported Mandibular Complete Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A03110220
Record Dates: First submitted 2021-12-15; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2021-12

CONDITIONS: Vertical Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned into two equal groups. Group I (control): patients who would be delivered mandibular implant overdenture retained by two RTX locator attachments using conventional loading protocol. Group II (study): patients who would be delivered mandibular overdenture retained by two RTx locator attachments using early loading protocol.
Who Masked: Participant, Outcomes Assessor
Masking Description: The selected patients were stratified according to age, gender, years of mandibular edentulism, number of old non-satisfactory dentures (baseline criteria, table 1). Patients were assigned to one of 2 groups using a balanced randomization procedure to ensure comparability between groups regarding baseline characters;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Group I (control): patients who would be delivered mandibular implant overdenture retained by two RTx locator attachments using conventional loading protocol
  Interventions: Procedure: surgical placement of long dental implants; Device: overdenture supported by RTX attachment system
- Study group (Active Comparator): Group II (study): patients who would be delivered mandibular overdenture retained by two RTx locator attachments using early loading protocol.
  Interventions: Procedure: surgical placement of long dental implants; Device: overdenture supported by RTX attachment system

INTERVENTIONS:
Procedure: surgical placement of long dental implants — Two interforaminal implants were placed in the canine region
Device: overdenture supported by RTX attachment system — Control group: Implants were loaded after three months by RTX supported overdenture study group: Implants were loaded after four weeks by RTX supported overdenture

SUMMARY:
This study was conducted to clinically and radiographically evaluate locator RTx attachments for two implant-supported mandibular overdenture using two loading protocols

DETAILED DESCRIPTION:
Thirty edentulous patients received two implants in the interformaninal region in the canine area . According to the loading protocol used for attaching mandibular overdenture, patients were randomly assigned into two equal groups. Group I (control): patients who would be delivered mandibular implant overdenture retained by two RTx locator attachments using conventional loading protocol. Group II (study): patients who would be delivered mandibular overdenture retained by two RTx locator attachments using early loading protocol. Peri-implant tissue health [Plaque (PL) and (GI) gingival scores, pocket depth (PD), and crestal bone loss (CBL)] were evaluated immediately after denture insertion (T0), 6 (T6), and 12 (T12) months after insertion.

ELIGIBILITY:
Inclusion Criteria:

* adequate bone quantity [class III -V according to Cawood and Howell in the interforaminal area of the mandible to receive 2 implants (4×13 mm)
* adequate restorative space [12-15 mm from the mucosa of the mandibular ridge to the occlusal plane, Class I according to Ahuja and Cagna for RTX supported implant overdenture.

Exclusion Criteria:

* systemic diseases that contraindicate implant placement
* bone metabolic diseases as diabetes mellitus
* irradiation of the head and neck region
* chemotherapy within the past 3 years
* smoking habits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | one year
  evaluations of crestal bone loss in mm around implants by digital periapical radiography
plaque score | one year
  evaluation of plaque accumulation around RTX attachments using scores.score 0; absence plaque , score 1; plaque only detected by a probe passing through the smooth marginal surface of the implant, score 2; plaque can be recognized by naked eye, and score 3; plenty of soft matter.
gingival index | one year
  evaluation of gingival bleeding around RTX attachments using scores.0; no bleeding when a periodontal probe is passed along the mucosal margin, 1;isolated bleeding spots visible, 2; blood forms a confluent red line on the mucosal margin, 3;heavy or profuse bleeding.
pocket depth | one year
  evaluation of pocket depth in mm around RTX attachments

CONTACTS AND LOCATIONS:
Locations (1):
- Christine Ibrahim, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No